CLINICAL TRIAL: NCT00138216
Title: A Phase I Study of Temozolomide, Oral Irinotecan, and Vincristine for Children With Refractory Solid Tumors
Brief Title: Temozolomide, Vincristine, and Irinotecan in Treating Young Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0414; COG-ADVL0414 (Other: Children's Oncology Group); CDR0000440069 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2023-10-02 (Actual); Status verified 2014-02

CONDITIONS: Brain and Central Nervous System Tumors; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood brain stem glioma; recurrent childhood brain tumor; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway and hypothalamic glioma; childhood oligodendroglioma; childhood craniopharyngioma; childhood choroid plexus tumor; childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; childhood central nervous system germ cell tumor; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood subependymal giant cell astrocytoma; childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma; Oligodendroglioma; Choroid Plexus Neoplasms; Rhabdoid Tumor | interventions — Irinotecan; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Irinotecan, temozolomide and vincristine sulfate (Experimental): see detailed description
  Interventions: Drug: irinotecan hydrochloride; Drug: temozolomide; Drug: vincristine sulfate

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: temozolomide
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, vincristine, and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan when given together with temozolomide and vincristine in treating young patients with refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of irinotecan when administered with temozolomide and vincristine in young patients with refractory solid tumors, including brain tumors.
* Determine the toxic effects of this regimen in these patients.
* Compare the toxic effects of this regimen in patients with low- vs high-risk UGT1A1 genotypes.
* Determine the pharmacokinetics of irinotecan in these patients.

Secondary

* Determine, preliminarily, the antitumor activity of this regimen in these patients.
* Correlate UGT1A1, UGT1A7, UGT1A9, and BCRP genotypes with the pharmacokinetics and pharmacodynamics of irinotecan and its metabolites in these patients.

OUTLINE: This is a multicenter, dose-escalation study of irinotecan. Patients are stratified according to UGT1A1 genotype (high-risk [7/7 or 6/7 genotype AND bilirubin ≥ 0.6 mg/dL] vs low-risk [absence of high-risk criteria]) if a high-risk patient experiences a dose-limiting toxicity (DLT).

Patients receive oral temozolomide on days 1-5 and oral irinotecan on days 1-5 and 8-12. Patients also receive vincristine IV over 1 minute on days 1 and 8. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT.

After completion of study treatment, patients are followed for 1 month and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* malignant solid tumor, including brain tumor, at original diagnosis or relapse

  * Refractory disease NOTE: *Histologic confirmation not required for intrinsic brain stem tumors
* Measurable or evaluable disease
* No known curative therapy OR therapy proven to prolong survival with an acceptable quality of life exists
* No known bone marrow metastases

PATIENT CHARACTERISTICS:

Age

* 1 to 21

Performance status

* Lansky 50-100% (for patients ≤ 10 years of age)
* Karnofsky 50-100% (for patients > 10 years of age)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (RBC transfusions allowed)

Hepatic

* ALT ≤ 110 U/L (upper limit of normal [ULN] for ALT is 45 U/L)
* Bilirubin ≤ 1.5 times ULN
* Albumin ≥ 2 g/dL

Renal

* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (for patients ≤ 5 years of age)
  * No greater than 1.0 mg/dL (for patients 6 to 10 years of age)
  * No greater than 1.2 mg/dL (for patients 11 to 15 years of age)
  * No greater than 1.5 mg/dL (for patients > 15 years of age)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Neurologic deficits in patients with CNS tumors must be stable for ≥ 1 week prior to study entry
* No uncontrolled infection
* No documented allergy to cephalosporins or dacarbazine

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* At least 3 months since prior stem cell transplantation or rescue without total-body irradiation

  * No evidence of active graft-versus-host disease
* At least 7 days since prior antineoplastic biologic agents
* At least 7 days since prior hematopoietic growth factors
* No concurrent biologic therapy or immunotherapy
* No concurrent prophylactic filgrastim (G-CSF) during the first course of study treatment

Chemotherapy

* Recovered from prior chemotherapy
* Prior temozolomide, vincristine, irinotecan, or topotecan allowed

  * No prior coadministration of temozolomide and irinotecan
  * No disease progression during treatment with either irinotecan or temozolomide
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas)
* No other concurrent chemotherapy

Endocrine therapy

* Patients with CNS tumors must be on a stable or decreasing dose of dexamethasone for ≥ 7 days prior to study entry

Radiotherapy

* Recovered from prior radiotherapy
* At least 6 months since prior total-body irradiation, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational drugs
* No other concurrent anticancer therapy
* No concurrent enzyme-inducing anticonvulsants, including any of the following:

  * Phenobarbital
  * Phenytoin
  * Carbamazepine
  * Oxcarbazepine
* No concurrent administration of any of the following:

  * Rifampin
  * Voriconazole
  * Itraconazole
  * Ketoconazole
  * Aprepitant
  * Hypericum perforatum (St. John's wort)
* No concurrent treatment for clostridium difficile infection

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) of oral irinotecan | length of study
  To estimate the maximum tolerated dose (MTD) of oral irinotecan administered on two different schedules together with fixed-dose temozolomide and vincristine in children with refractory solid tumors or brain tumors

SECONDARY OUTCOMES:
To preliminarily define the antitumor activity | Length of study
  To preliminarily define the antitumor activity of this drug combination within the confines of a Phase 1 study.

CONTACTS AND LOCATIONS:
Overall Officials: Lars M. Wagner, MD, Study Chair — Children's Hospital Medical Center, Cincinnati; John P. Perentesis, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (18):
- United States (16):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Stanford Cancer Center, Stanford, California
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Wagner LM, Perentesis JP, Reid JM, Ames MM, Safgren SL, Nelson MD Jr, Ingle AM, Blaney SM, Adamson PC. Phase I trial of two schedules of vincristine, oral irinotecan, and temozolomide (VOIT) for children with relapsed or refractory solid tumors: a Children's Oncology Group phase I consortium study. Pediatr Blood Cancer. 2010 Apr;54(4):538-45. doi: 10.1002/pbc.22407. PMID 20049936